CLINICAL TRIAL: NCT00315705
Title: A Phase 1/2 Dose-Escalation Study of Clofarabine in Combination With Etoposide and Cyclophosphamide in Pediatric Patients With Refractory or Relapsed Acute Leukemias.
Brief Title: A Study of Clofarabine in Combination With Etoposide and Cyclophosphamide in Children With Acute Leukemias.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO21800205
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myelogenous Leukemia; Relapsed Leukemia
Keywords: clofarabine; acute leukemia; ALL; AML; clolar; CLO218
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia | interventions — Clofarabine; Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clofarabine, etoposide, cyclophosphamide (Experimental): Phase 1: escalating dosage of the three drugs delivered intravenously. Clofarabine dosage from 20-40 mg/m^2, etoposide dosage from 75-100 mg/m^2, cyclophosphamide dosage from 340-440 mg/m^2.
  Phase 2: The recommended phase 2 doses (RP2D) were clofarabine 40 mg/m^2, etoposide 100 mg/m^2 and cyclophosphamide 440 mg/m^2 delivered intravenously
  Interventions: Drug: clofarabine; Drug: Etoposide; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: clofarabine — Clofarabine 20-40 mg/m²/day 2 hour intravenous (IV) infusion daily for 5 days of a 28 day cycle as the first of the three IV interventions administered. Maximum of 8 cycles given in both the phase 1 and phase 2 study periods.
  Other Names: Clolar; Evoltra
Drug: Etoposide — Etoposide 75-100 mg/m²/day 2 hour intravenous (IV) infusion daily for 5 days of a 28 day cycle following clofarabine therapy. Maximum of 8 cycles given in both the phase 1 and phase 2 study periods.
  Other Names: Eposin
Drug: Cyclophosphamide — Cyclophosphamide 340-440 mg/m²/day as 30-60 minute intravenous (IV) infusion daily for 5 days of a 28 day cycle following the other two interventions. Maximum of 8 cycles given in both the phase 1 and phase 2 study periods.
  Other Names: Endoxan; Revimmune; Cytoxan

SUMMARY:
Clofarabine (injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed or refractory acute lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens. This use is based on the induction of complete responses. Randomized trials demonstrating increased survival or other clinical benefit have not been conducted.

The purpose of the phase 1 portion of this study was to determine if clofarabine added to a combination of etoposide and cyclophosphamide is safe in children with relapsed or refractory acute lymphoblastic leukemia (ALL) or acute myelogenous leukemia (AML). The purpose of the phase 2 portion of the study was to measure the effectiveness of the combination therapy in children with ALL.

ELIGIBILITY:
Inclusion Criteria:

* NOTE: the following eligibility criteria were applicable to acute lymphoblastic leukemia (ALL) and acute myelogenous leukemia (AML) patients for the Phase 1 portion of this study, and to ALL patients for the Phase 2 portion of the study (only ALL patients were allowed in the Phase 2 portion of the study).
* ALL with > 25% blasts in bone marrow; AML with ≥ 5% blasts in bone marrow; ALL and AML patients may have extramedullary disease
* Karnofsky Performance Status ≥ 50 for patients > 10 years old; Lansky Performance Status ≥ 50 for patients ≤ 10 years old
* Prior therapy: AML: 1-2 prior induction regimens and ≤ 1 hematopoietic stem cell transplant (HSCT); ALL: 1-3 prior induction regimens
* Adequate liver, renal, pancreatic, and cardiac function
* Have received no prior HSCT (study amended in Phase 2 to exclude patients with prior HSCT)

Exclusion Criteria:

* NOTE: the following eligibility criteria were applicable to ALL and AML patients for the Phase 1 portion of this study, and to ALL patients for the Phase 2 portion of the study (only ALL patients were allowed in the Phase 2 portion of the study).
* Burkitt's leukemia
* Previous treatment with clofarabine
* Uncontrolled systemic fungal, bacterial or other infection and 48 hrs negative blood cultures required for patients with a history of fever within 3 days of enrollment
* Active CNS involvement (i.e., should be CNS1 or CNS2)
* Inadequate time since last therapy: ≤ 14 days since last cytotoxic chemotherapy; ≤ 7 days since last biologic therapy; ≤ 14 days since last monoclonal antibody therapy
* Have received prior HSCT (study amended in Phase 2 to exclude patients with prior HSCT)
* Pregnant or lactating
* Have tested positive for hepatitis B or hepatitis C infection or history of cirrhosis

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (13):
- United States (13):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Memorial Hospital, Chicago, Illinois
  - St. Vincent Children's Hospital, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York School of Medicine, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Hijiya N, Thomson B, Isakoff MS, Silverman LB, Steinherz PG, Borowitz MJ, Kadota R, Cooper T, Shen V, Dahl G, Thottassery JV, Jeha S, Maloney K, Paul JA, Barry E, Carroll WL, Gaynon PS. Phase 2 trial of clofarabine in combination with etoposide and cyclophosphamide in pediatric patients with refractory or relapsed acute lymphoblastic leukemia. Blood. 2011 Dec 1;118(23):6043-9. doi: 10.1182/blood-2011-08-374710. Epub 2011 Oct 3. PMID 21967976

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine, Etoposide, Cyclophosphamide: Phase 1: escalating dosage of the three drugs delivered intravenously. Clofarabine dosage from 20-40 mg/m^2, etoposide dosage from 75-100 mg/m^2, cyclophosphamide dosage from 340-440 mg/m^2.> Phase 2: The recommended phase 2 doses (RP2D) were clofarabine 40 mg/m^2, etoposide 100 mg/m^2 and cyclophosphamide 440 mg/m^2 delivered intravenously
Period: Phase 1
Arm/Group | Clofarabine, Etoposide, Cyclophosphamide
Started | 25
Completed | 0 (No Phase 1 participants completed the treatment period (i.e. all 8 cycles and follow-up))
Not Completed | 25
Not completed — Refused further treatment | 1
Not completed — Failure to achieve response | 8
Not completed — Disease relapse | 4
Not completed — Scheduled for transplant | 9
Not completed — Death | 3
Period: Phase 2
Arm/Group | Clofarabine, Etoposide, Cyclophosphamide
Started | 25 (Phase 1 and phase 2 are separate populations)
Completed | 0 (No Phase 2 participants completed the treatment period (i.e. all 8 cycles and follow-up))
Not Completed | 25
Not completed — Physician Decision | 4
Not completed — Adverse Event | 1
Not completed — Failure to achieve response | 3
Not completed — Disease relapse | 1
Not completed — Scheduled for transplant | 8
Not completed — Other | 1
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Clofarabine, Etoposide, Cyclophosphamide: Phase 1: escalating dosage of the three drugs delivered intravenously. Clofarabine dosage from 20-40 mg/m^2, etoposide dosage from 75-100 mg/m^2, cyclophosphamide dosage from 340-440 mg/m^2.
- Phase 2: Clofarabine, Etoposide, Cyclophosphamide: Phase 2: The recommended phase 2 doses (RP2D) were clofarabine 40 mg/m^2, etoposide 100 mg/m^2 and cyclophosphamide 440 mg/m^2 delivered intravenously
- Total: Total of all reporting groups
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide | Phase 2: Clofarabine, Etoposide, Cyclophosphamide | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — The two study phases were not designed to be reported in the aggregate.
  years | 9.1 (5.03) | 13.2 (5.25) | 11.2 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants] — The two study phases were not designed to be reported in the aggregate.
  Participants
    Female | 10 | 9 | 19
    Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The two study phases were not designed to be reported in the aggregate.
  Participants
    Hispanic or Latino | 5 | 10 | 15
    Not Hispanic or Latino | 20 | 15 | 35
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The two study phases were not designed to be reported in the aggregate.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 2 | 6
    White | 16 | 12 | 28
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 2 | 8 | 10
Percent Leukemic Blast Cells [Mean (Standard Deviation); unit: percentage of total blast cells] — Percent of leukemic blast cells based on bone marrow aspirate. The two study phases were not designed to be reported in the aggregate.
  percentage of total blast cells | 66.8 (24.85) | 69.52 (23.566) | 68.16 (24.008)
Absolute Neutrophil Counts [Mean (Standard Deviation); unit: 10^9/L] — The two study phases were not designed to be reported in the aggregate.
  10^9/L | 1.93828 (3.049992) | 1.9280 (1.708126) | 1.93325 (2.459536)
White Blood Cell Counts [Mean (Standard Deviation); unit: 10^9/L] — The two study phases were not designed to be reported in the aggregate.
  10^9/L | 8.323 (9.1305) | 12.171 (23.0150) | 10.247 (17.4370)
Immunophenotype [Number; unit: participants] — Applies to acute lymphoblastic leukemic (ALL) participants only. Acute myelogenous leukemic (AML) participants are not included. The two study phases were not designed to be reported in the aggregate.
  participants
    B cell | 13 | 21 | 34
    T cell | 5 | 1 | 6
    Unknown | 2 | 3 | 5
    not included (AML participants) | 5 | 0 | 5
Count of Previous Anti-Leukemic (non-transplant) Treatment Regimens [Number; unit: participants] — The two study phases were not designed to be reported in the aggregate.
  participants
    1 regimen | 4 | 4 | 8
    2 regimens | 18 | 14 | 32
    3 regimens | 3 | 7 | 10
Participants with Previous Anti-Leukemic Transplant Regimens [Number; unit: participants] — The two study phases were not designed to be reported in the aggregate.
  participants
    Transplants | 4 | 4 | 8
    No transplants | 21 | 21 | 42
Participants Who Were Refractory to the Most Recent Previous Anti-Leukemic Treatment [Number; unit: participants] — The answer "Yes" indicates the number of participants who were refractory (unresponsive) to the most recent anti-leukemic treatment. The answer "No" represents participants who were not refractory. The two study phases were not designed to be reported in the aggregate.
  participants
    Yes | 7 | 15 | 22
    No | 18 | 10 | 28
Participant Rating Using the Karnofsky/Lansky Performance Status Scale [Number; unit: participants] — Baseline performance was rating using either the Karnofsky Performance Scale for participants greater than 10 years old, or the Lansky Performance Scale for participants 10 years or younger. Both scales range from 0-100 with 0 indicating dead or unresponsive and 100 indicating normal performance. The two study phases were not designed to be reported in the aggregate.
  participants
    50 | 0 | 2 | 2
    60 | 0 | 2 | 2
    70 | 1 | 2 | 3
    80 | 5 | 3 | 8
    90 | 7 | 6 | 13
    100 | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) in Phase 1
Description: The MTD was to be the highest dose level of clofarabine in combination with etoposide and cyclophosphamide that caused <= 1 of 6 participants to experience a dose limiting toxicity (DLT) with the next higher dose level having at least 2 of 3 or 2 of 6 participants experiencing a DLT. The MTD would be used as the recommended phase 2 dose (RP2D). If the MTD could not be determined, then the target dose of clofarabine 40 mg/m^2, etoposide 100 mg/m^2 and cyclophosphamide 440 mg/m^2 as taken by Cohort 5 was to become the RP2D.
  The rating scale used is 0 = not the MTD, 1 = the MTD.
Time Frame: Up to Day 42 (Phase 1 portion of study)
Population: All phase 1 participants
Measure: Number; unit: units on a scale
Groups:
- Phase 1 - Cohort 1: Participants were treated with clofarabine 20 mg/m^2, etoposide 75 mg/m^2, and cyclophosphamide 340 mg/m^2.
- Phase 1 - Cohort 2: Participants were treated with clofarabine 20 mg/m^2, etoposide 75 mg/m^2, and cyclophosphamide 440 mg/m^2.
- Phase 1 - Cohort 3: Participants were treated with clofarabine 20 mg/m^2, etoposide 100 mg/m^2, and cyclophosphamide 440 mg/m^2.
- Phase 1 - Cohort 4: Participants were treated with clofarabine 30 mg/m^2, etoposide 100 mg/m^2, and cyclophosphamide 440 mg/m^2.
- Phase 1 - Cohort 5: Participants were treated with clofarabine 40 mg/m^2, etoposide 100 mg/m^2, and cyclophosphamide 440 mg/m^2.
Arm/Group | Phase 1 - Cohort 1 | Phase 1 - Cohort 2 | Phase 1 - Cohort 3 | Phase 1 - Cohort 4 | Phase 1 - Cohort 5
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 6
units on a scale | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Participants With Dose Limiting Toxicity in Phase 1
Description: The number of participants in each cohort that had dose limiting toxicity is summarized. Toxicities were reviewed by an independent Data Safety Monitoring Board (DSMB) who determined if additional participants should be added to the cohort and the criteria for escalating to the next cohort.
Time Frame: Up to Day 42 (Phase 1 portion of study)
Population: All phase 1 participants
Measure: Number; unit: participants
Arm/Group | Phase 1 - Cohort 1 | Phase 1 - Cohort 2 | Phase 1 - Cohort 3 | Phase 1 - Cohort 4 | Phase 1 - Cohort 5
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 6
participants | 0 | 0 | 0 | 1 | 1

3. Secondary Outcome: Summary of Participants With Adverse Events (AEs) in Phase 1
Description: Number of participants with AEs that occurred during treatment and follow-up period (45 days after last cycle). Drug-related AEs and SAEs were followed until resolved or mutually agreed by the investigator and Genzyme to discontinue reporting. AEs were classified by the investigator according to severity (graded using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 3.0) and relationship to study drug. The severity scale is:> Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death related to AE
Time Frame: Up to 9.5 months (Phase 1 portion of study)
Population: All phase 1 participants
Measure: Number; unit: participants
Arm/Group | Phase 1 - Cohort 1 | Phase 1 - Cohort 2 | Phase 1 - Cohort 3 | Phase 1 - Cohort 4 | Phase 1 - Cohort 5
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 6
participants
  At least one AE | 3 | 3 | 3 | 10 | 6
  At least one AE related to clofarabine | 3 | 3 | 3 | 10 | 6
  At least one serious AE | 3 | 3 | 3 | 9 | 6
  At least one serious AE related to clofarabine | 3 | 2 | 3 | 9 | 5
  Discontinued study due to AE | 0 | 0 | 0 | 0 | 0
  Died | 3 | 1 | 3 | 9 | 5
  AE with the worst grade of: 1 | 0 | 0 | 0 | 0 | 0
  AE with the worst grade of: 2 | 0 | 0 | 0 | 0 | 0
  AE with the worst grade of: 3 | 2 | 1 | 1 | 3 | 3
  AE with the worst grade of: 4 | 1 | 1 | 2 | 5 | 2
  AE with the worst grade of: 5 | 0 | 1 | 0 | 2 | 1

4. Secondary Outcome: Percentage of Participants Achieving A Response Over the First Two Treatment Cycles in Phase 1
Description: Response categories 1) complete remission (CR): without circulating blasts or extramedullary disease, bone marrow (BM) with <5% blasts, and platelet (plt)/ANC recovery: ALL ≥75/ ≥0.75 [x 10^9/L]; AML ≥100/ ≥1.0 [x 10^9/L] 2) CR in absence of plt recovery (CRp): ALL plt ≥20 to <75 x 10^9/L; AML plt ≥20 to <100 x 10^9/L 3) partial remission (PR): no circulating blasts, appearance of normal hematopoietic progenitors, and either a BM with ≥5% and ≤25% blasts with recovery of plts/ANC or a BM with <5% blasts not meeting CR/CRp definition 4) Overall remission (OR): CR+CRp 5) Any response: CR+CRp+PR.
Time Frame: Approximately 2 months (Phase 1 portion of study)
Population: All phase 1 participants
Measure: Number; unit: percentage of total participants
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
percentage of total participants
  Complete remission (CR) | 40
  Complete remission/absence total platelet recovery | 24
  Partial remission (PR) | 0
  Overall remission (OR) | 64
  Any response (CR+CRp+PR) | 64

5. Secondary Outcome: Time to Remission for Participants Who Had a Response in Phase 1
Description: The weeks between start of intervention and remission as assessed by the investigator in Phase 1. Participants who had a complete remission (CR) or complete remission with the absence of total platelet recovery (CRp) are included.
Time Frame: up to 8 weeks (Phase 1 portion of study)
Population: Participants in phase 1 who had an overall remission.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 16
weeks | 4.96 (1.912)

6. Secondary Outcome: Kaplan Meier Estimate of Duration of Remission (DOR) for Participants Who Achieved Overall Remission (OR) in Phase 1
Description: Duration of response is the time from the first objective measurement of complete response (CR) or complete response with the absence of total platelet recovery (CRp) to the date of first objective documentation of disease relapse or death due to any cause, plus one day. For summary purposes, results are presented as weeks.
Time Frame: Up to 2 years (Phase 1 portion of study)
Population: Phase 1 participants who achieved overall remission. Data are censored at date of last known follow-up visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 16
weeks | 18.2 [12.9 to 35.0]

7. Secondary Outcome: Kaplan Meier Estimates of Event-free Survival (EFS) for Participants in Phase 1
Description: Event-free survival (EFS) is defined as the time from date of first administration of study interventions until the earliest of the following: date of death or date of first response assessment confirming relapse or date of final response assessment which fails to confirm response, plus one day. For summary purposes, results are presented as weeks.
Time Frame: Up to 2 years (Phase 1 portion of study)
Population: All phase 1 participants. Data are censored at date of last known follow-up visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
weeks | 19.3 [12.7 to 27.1]

8. Secondary Outcome: Number of Participants With 4-month Event Free Survival in Phase 1
Description: Number of participants with event-free survival at four months post first dose of therapy. A participant is considered event-free if at month 4 they have not died or had a response assessment confirming a relapse.
Time Frame: 4 months (Phase I portion of study)
Population: All participants
Measure: Number; unit: participants
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
participants | 13

9. Secondary Outcome: Kaplan Meier Estimates of Overall Survival (OS) for Participants in Phase 1
Description: Overall survival is defined as the time from date of first administration of study interventions until date of death, plus one day. For summary purposes, results are presented as weeks.
Time Frame: Up to 2 years (Phase 1 portion of study)
Population: All phase 1 participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 1: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
weeks | 27.1 [18.3 to 42.9]

10. Primary Outcome: Percentage of Participants Achieving A Response Over the First Two Treatment Cycles in Phase 2
Description: Response categories 1) complete remission (CR): without circulating blasts or extramedullary disease, bone marrow (BM) with <5% blasts, and platelet (plt)/ANC recovery: ≥75/ ≥0.75 [x 10^9/L] 2) CR in absence of plt recovery (CRp): plt ≥20 to <75 x 10^9/L 3) partial remission (PR): no circulating blasts, appearance of normal hematopoietic progenitors, and either a BM with ≥5% and ≤25% blasts with recovery of plts/ANC or a BM with <5% blasts not meeting CR/CRp definition 4) Overall remission (OR): CR+CRp 5) Any response: CR+CRp+PR.
Time Frame: Approximately 28-56 days (Phase 2 portion of study)
Population: All phase 2 participants
Measure: Number; unit: percentage of total participants
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
percentage of total participants
  Complete remission (CR) | 28
  Complete remission/absence total platelet recovery | 16
  Partial remission (PR) | 12
  Overall remission (OR) | 44
  Any response (CR+CRp+PR) | 56

11. Secondary Outcome: Summary of Participants With Adverse Events (AEs) in Phase 2
Description: as for outcome 3
Time Frame: Up to 9.5 months (Phase 2 portion of study)
Population: All phase 2 participants
Measure: Number; unit: participants
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
participants
  At least one AE | 25
  At least one AE related to clofarabine | 25
  At least one serious AE | 21
  At least one serious AE related to clofarabine | 20
  Discontinued study due to AE | 1
  Died | 16
  AE with the worst grade of: 1 | 0
  AE with the worst grade of: 2 | 0
  AE with the worst grade of: 3 | 1
  AE with the worst grade of: 4 | 16
  AE with the worst grade of: 5 | 8

12. Secondary Outcome: Time to Remission for Participants Who Had a Response in Phase 2
Description: The weeks between start of intervention and remission as assessed by the investigator in Phase 2. Participants who had a complete remission (CR) or complete remission with the absence of total platelet recovery (CRp) are included.
Time Frame: up to 8 weeks (Phase 2 portion of study)
Population: Participants in phase 2 who had an overall remission.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 11
weeks | 4.84 (2.092)

13. Secondary Outcome: Kaplan Meier Estimate of Duration of Remission (DOR) for Participants Who Achieved Overall Remission (OR) in Phase 2
Description: as for outcome 6
Time Frame: Up to 2 years (Phase 2 portion of study)
Population: Phase 2 participants who achieved overall remission. Data are censored at date of last known follow-up visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 11
weeks | 67.3 [13.4 to NA] — NA = not estimable because values are mostly censored. Participants with longer DORs have not relapsed, progressed, or died, therefore the upper confidence limit cannot be estimated.

14. Secondary Outcome: Kaplan Meier Estimates of Event-free Survival (EFS) for Participants in Phase 2
Description: as for outcome 7
Time Frame: Up to 2 years (Phase 2 portion of study)
Population: All phase 2 participants. Data are censored at date of last known follow-up visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
weeks | 10.7 [6.7 to 73.9]

15. Secondary Outcome: Number of Participants With 4-month Event Free Survival in Phase 2
Description: as for outcome 8
Time Frame: 4 months (Phase 2 portion of study)
Population: All participants
Measure: Number; unit: participants
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
participants | 11

16. Secondary Outcome: Kaplan Meier Estimates of Overall Survival (OS) for Participants in Phase 2
Description: as for outcome 9
Time Frame: Up to 2 years (Phase 2 portion of study)
Population: All phase 2 participants. Data are censored at date of last known follow-up visit.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Number analyzed (Participants) | 25
weeks | 10.7 [8.1 to 38.6]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse experiences collected in Phase 1 from day 1 up to 9.5 months. Phase 2 also lasted up to 9.5 months and started after Phase 1.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of adverse event tables.
Groups:
- Phase 1 - Total: All participants from Cohorts 1-5 in Phase 1
Arm/Group | Phase 1 - Cohort 1 | Phase 1 - Cohort 2 | Phase 1 - Cohort 3 | Phase 1 - Cohort 4 | Phase 1 - Cohort 5 | Phase 1 - Total | Phase 2: Clofarabine, Etoposide, Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/10 | 6/6 | 24/25 | 21/25
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 10/10 | 6/6 | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Cohort 1 (N=3) | Phase 1 - Cohort 2 (N=3) | Phase 1 - Cohort 3 (N=3) | Phase 1 - Cohort 4 (N=10) | Phase 1 - Cohort 5 (N=6) | Phase 1 - Total (N=25) | Phase 2: Clofarabine, Etoposide, Cyclophosphamide (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 7 | 3 | 17 | 15
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2 | 5 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intracardiac mass (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Trichiasis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Caecitis (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 3 | 2 | 0 | 6 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BK virus infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 3 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Central nervous system infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cerebral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 3 | 2
Ear infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 2
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Meningitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Otitis media bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 3 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Viraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | 1
Polyomavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Venoocclusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Cohort 1 (N=3) | Phase 1 - Cohort 2 (N=3) | Phase 1 - Cohort 3 (N=3) | Phase 1 - Cohort 4 (N=10) | Phase 1 - Cohort 5 (N=6) | Phase 1 - Total (N=25) | Phase 2: Clofarabine, Etoposide, Cyclophosphamide (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1 | 2 | 7 | 16
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 13
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 5 | 3 | 11 | 16
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 3 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 3 | 2 | 6 | 7
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 1 | 1 | 4 | 0
Mixed deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0
Ectropion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 9 | 2 | 13 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 1 | 9 | 5
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 7 | 5 | 17 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 9 | 5 | 21 | 20
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Oral pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pancreatic atrophy (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 3
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 3
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3 | 9 | 6 | 22 | 22
Application site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 2
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 2 | 0 | 1 | 4 | 4
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 2 | 2 | 6 | 2
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 2 | 3 | 5 | 6
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2
Pneumatosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 1 | 7 | 5 | 15 | 13
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 3 | 0 | 4 | 5
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0 | 3 | 6
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BK virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 3 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2 | 2
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster multi-dermatomal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Keratitis herpetic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 3
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2 | 4 | 3
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 2 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 3 | 8
Antimicrobial susceptibility test sensitive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 2 | 11
Bacterial test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Coagulation test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Culture stool positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fibrin d dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 2 | 5
Occult blood positive (Investigations) | 0 | 0 | 1 | 0 | 1 | 2 | 1
Polyomavirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Specific gravity urine abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Specific gravity urine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Urine ketone body (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 5 | 4 | 12 | 15
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 3 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 3 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 6 | 1 | 11 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 1 | 5 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 2 | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 8
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 4 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 5 | 3 | 11 | 6
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 4 | 1 | 7 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 7 | 4 | 14 | 9
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 2 | 4 | 2 | 10 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1 | 4 | 3
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Social avoidant behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 2 | 4 | 6
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Kidney enlargement (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3 | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 1 | 7 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2 | 5 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 3 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 2
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 6 | 4
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1 | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 6
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 5 | 2 | 8 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 6 | 4 | 14 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2 | 5 | 2 | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.